CLINICAL TRIAL: NCT02836288
Title: A Randomized, Double Blind, Feasibility Study of Oral Ketamine Versus Placebo for Treating Depression in Patients With Cancer
Brief Title: Study of Oral Ketamine Versus Placebo for Treating Depression in Patients Undergoing Treatment for Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Scott A. Irwin, MD, PhD (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor-Investigator, Scott A. Irwin, MD, PhD, Associate Professor, Psychiatry & Behavioral Neurosciences, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IIT2015-23-IRWIN-KETTREAT
Record Dates: First submitted 2016-07-14; First posted 2016-07-19 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Cancer; Depression
Keywords: Ketamine; Treatment of Depression
MeSH Terms: conditions — Neoplasms; Depression | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Ketamine (Experimental): Oral ketamine 1.0 mg/kg mixed with syrup
  Interventions: Drug: Ketamine
- Placebo (Placebo Comparator): Oral placebo (syrup)
  Interventions: Other: Placebo
- Ketamine after placebo (Experimental): Optional oral Ketamine 1.0 mg/kg mixed with syrup for patients on placebo arm after 12 week treatment is completed.
  Interventions: Drug: Ketamine; Other: Placebo

INTERVENTIONS:
Drug: Ketamine — Ketamine 1.0 mg/kg mixed with syrup will be given by mouth once a day for 12 weeks.
  Other Names: Ketalar
  Arms: Ketamine; Ketamine after placebo
Other: Placebo — Placebo syrup will be given by mouth once a day for 12 weeks.
  Arms: Ketamine after placebo; Placebo

SUMMARY:
The primary purpose of this study is to see if it is safe to give patients with cancer a low dose of the FDA approved anesthetic drug ketamine at the same time they receive radiation, chemotherapy, and/or surgery for their cancer treatment to treat depression and its effects. Researchers would also like to see if giving ketamine at the same time as cancer treatment is practical and reasonably acceptable to the patient.

Depression has many negative consequences for outcomes in those with cancer. It causes delayed treatments, increases in hospital lengths of stay, decreases in treatment adherence, poorer self-care, and decreased quality of life, even at 3 years post treatment. The presence of depression is the number one predictor of incomplete treatment and difficulty with rehabilitation. Therefore, investigators would also like to see if it is feasible to give patients ketamine during their routine cancer treatment treat depression and its negative effects on cancer treatment outcomes, and also help with anxiety, pain, and quality of life. The study will also use a placebo to compare to the good and/or bad effects of ketamine. A placebo is not an active drug and it will be look the same as ketamine, as a liquid to be taken by mouth.

Ketamine is approved by the U.S. Food and Drug Administration (FDA) as a general anesthetic by itself for some diagnostic and surgical procedures or combined with other general anesthetic agents. It has also been shown to reduce cancer pain. Ketamine is considered experimental in this study because it is not approved by the FDA for the treatment of depression.

DETAILED DESCRIPTION:
This is a prospective, single center, double blind, randomized, two-arm feasibility study of oral ketamine versus placebo for the treatment of depression in depressed patients with cancer undergoing curative intent cancer therapy. Approximately 20 patients with cancer about to undergo cancer therapy will be randomized 1:1 to receive study treatment with one of the following regimens:

Arm A: nightly oral administration of 1.0 mg/kg ketamine Arm B: nightly oral administration of placebo (after completion of Arm B, patients will have the option to receive a nightly oral administration of 1.0 mg/kg ketamine and follow study procedures over again)

Consenting patients will undergo screening procedures, and if eligible, a baseline interview and brief questionnaires regarding depression, mental and emotional health, and quality of life assessments.

Study treatment will be administered for 12 weeks unless the patient experiences unacceptable toxicities, exhibits moderate to severe depressive symptoms, or withdraws consent. Patients on the placebo treatment arm will have the option to receive ketamine and follow all study procedures over again with the ketamine drug after completion of the placebo treatment.

Patients will be asked to complete psychosocial measurements every two weeks while on study treatment and monthly during a five-month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent.
* Subject receiving or within twelve weeks of having received curative intent cancer treatment with radiation and/or chemotherapy
* Age ≥ 18 years.
* Has moderate to severe depression according to Quick Inventory of Depressive Symptomatology-Self Rated 16 (QIDS-SR-16) scores of ≥ 11 AND a Hospital Anxiety and Depression Scale (HADS) Depression subscale score of ≥ 8.
* Documented adequate liver function within the screening period as defined by:
* ALT < 5 X institutional upper limit of normal (ULN)
* AST < 5 X institutional ULN
* Total bilirubin < 5 X institutional ULN
* Both men and women of all races and ethnic groups are eligible for this trial.
* Use of other antidepressants is permitted if dose has been the same for at least 12 weeks prior to study entry and still meet inclusion #4.
* Women of child-bearing potential and men with partners of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating and the study physician immediately. Urine pregnancy testing will be done throughout the trial for women of childbearing potential.
* Must read and understand English fluently.

Exclusion Criteria:

* Receiving another investigational agent on a clinical trial that prohibits participation in other studies of investigational agents.
* Meets MINI International Neuropsychiatric Interview (MINI Plus), criteria for diagnoses of schizophrenia, bipolar illness, delirium or psychosis.
* Has high Suicidal Risk Assessment (SRA) scores ≥ 10.
* Use of monoamine oxidase inhibitors within 14 days of study entry.
* History of allergic reactions or hypersensitivity to ketamine.
* Documented history of severe cardiac insufficiency (NYHA III or IV), with uncontrolled and/or unstable cardiac or coronary artery disease.
* Documented history of significant tachyarrhythmia, severe angina, or myocardial ischemia
* Documented history of poorly controlled hypertension (Systolic Blood Pressure > 180 mmHG or Diastolic Blood Pressure > 100 mmHG), with or without antihypertensives.
* If a woman is or becomes pregnant or is nursing at any time before or during the treatment period, she will be excluded from the study.
* Score of ≥ 8 on the WHO Alcohol Use Disorders Identification Test (AUDIT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-12-20 (Actual); Primary Completion 2018-05-29 (Actual); Study Completion 2018-05-29 (Actual)

PRIMARY OUTCOMES:
Proportion of patients pre-screened that were potentially eligible for study participation. | 24 months
Proportion of patients that were potentially eligible who were approached. | 24 months
Proportion of approached patients that decline study participation and why. | 24 months
Proportion of approached patients that agreed to participate | 24 months
Proportion of approached that were randomized. | 24 months
Proportions of patients discontinuing prematurely from study treatment for any reason, including side effects attributed to ketamine or side effects attributed to placebo, documenting reasons for dropout. | 24 months
Proportion of patients evaluable. | 24 months

SECONDARY OUTCOMES:
Adverse events related to study treatment. | 10 months
Patient-reported Frequency, Intensity and Burden of Side Effects (FIBSER) scores. | 10 months
Treatment expectancy and satisfaction as measured by the credibility/expectancy questionnaire (CEQ). | 10 months

OTHER OUTCOMES:
Changes in scores for QIDS-SR-16 questionnaire. | 10 months
Changes in scores for Pain VAS questionnaire. | 10 months
Changes in scores for HADS questionnaire. | 10 months
Changes in scores for UW-QOL questionnaire. | 10 months
Changes in scores for SRA questionnaire. | 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Scott Irwin, MD, PhD, Principal Investigator — Cedars-Sinal Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States